CLINICAL TRIAL: NCT07093047
Title: A National Survey on the Perceived Effects of Italian Law 219/2017 in Pediatric Intensive Care Units
Brief Title: Effects of Italian Law 219/2017 in Pediatric Intensive Care Units
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: PES-219-PICU
Record Dates: First submitted 2025-07-03; First posted 2025-07-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Refusal of Treatment
MeSH Terms: conditions — Treatment Refusal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare personnel: Healthcare personnel employed in pediatric intensive care units
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — Participants are required to complete a survey collecting anonymous data

SUMMARY:
This study aims to investigate pediatric intensive care providers' knowledge, perceptions, and experiences with Law 219/2017 by means of a national multicentric non-interventional cross-sectional study.

DETAILED DESCRIPTION:
In Italy in January 2018, Law 219/2017 came into effect after years of discussion regarding the possibility of refusing potentially life-saving health treatments, with its general principles being respect of life, human dignity, and personal self-determination, and introducing the concept of Advance Care Planning, the possibility for the patient to refuse medical treatment stating also that the patient cannot demand health treatments contrary to the law, professional ethics or good clinical-care practices letting the physician protected by the law in not providing interventions that he/she judges contrary to the patient's best health interest.

This study aims to investigate pediatric intensive care providers' knowledge, perceptions, and experiences with Law 219/2017 by means of a national multicentric non-interventional cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare personnel employed in a pediatric intensive care units

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare personnel employed in a pediatric intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Knowledge of the Italian Law 219/2017 | Through study completion, an average of three months
  The level of knowledge of the Italian law 219/2017, will be assessed through a survey developed drafting questions and answers by a multiprofessional panel of international experts in PICU, Bioethics, and research methodology. This survey contains questions on the law and also personal reflections on the choices made by healthcare professionals in the case studies included.
  The questions will not be given a score, the data analysis will be purely qualitative.
Experience about the application of the Italian Law 219/2017 | Through study completion, an average of three months
  The questions, which were constructed by a multidisciplinary team, contain a section to explore the personal experience of the respondents during their shifts in intensive care.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Martinato, PhD, Principal Investigator — University of Padova
Locations (3):
- Italy (3):
  - Ospedale Sant'Orsola Malpighi, Bologna
  - Ospedale Gaslini, Genova
  - Università di Torino, Torino

IPD SHARING:
Plan to Share IPD: Undecided